CLINICAL TRIAL: NCT05753163
Title: Hepatic Arterial Infusion Chemotherapy Combined With Sintilimab and Regorafenib as Adjuvant Therapy for Colorectal Liver Metastasis Patients With a High Risk of Recurrent: a Single-arm, Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Director of Hepatic Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-GWK-001
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Liver Metastasis
MeSH Terms: interventions — sintilimab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Combination Product: HAIC-FOLFOX combined with Sintilimab and Regorafenib

INTERVENTIONS:
Combination Product: HAIC-FOLFOX combined with Sintilimab and Regorafenib — HAIC (FOLFOX: oxaliplatin 85mg/m2, 5- fluorouracil 2500mg/m2, calcium folinate 400mg/m2) was given every 4-6 weeks for 2-4 cycles depending on pts' health status, in combination with Sintilimab (200mg, iv, d1) and regorafenib (80mg, po, d1-21) every 3 weeks for up to 6 months .

SUMMARY:
Pts with histologically confirmed CRLM and whose CRS >2 were enrolled into this single-arm, phase II study. The critical enrollment criteria were that Subjects had completely resected Primary lesion and liver metastases and had no evidence of extrahepatic disease. After hepatectomy， HAIC (FOLFOX: oxaliplatin 85mg/m2, 5- fluorouracil 2500mg/m2, calcium folinate 400mg/m2) was given every 4-6 weeks for 2-4 cycles depending on pts' health status, in combination with Sintilimab (200mg, iv, d1) and regorafenib (80mg, po, d1-21) every 3 weeks for up to 6 months. The primary endpoint was 1-year recurrence-free survival (RFS) and secondary endpoints included RFS, overall survival (OS), safety, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years， men or women who are not pregnant；
2. ECOG PS 0/1 evaluated 14 days before enrollment, and expected survival >12 months after liver resection;
3. Liver function: Child-Pugh score Class A or ≤7 Class B；
4. Patients with histologically- or clinically-confirmed CRLM（TxNxM1）and CRS>2；
5. Patients had completely resected Primary lesions and liver metastases as well as no evidence of extrahepatic disease；
6. No complications such as bleeding, jaundice, infection, abdominal pleural effusion, obstruction and perforation were observed within 7 days (including 7 days) before the screening. The subjects recovered well after surgery, the surgical incision healed well, the stitches were removed, and the drainage tube was removed;
7. Preoperative chemoradiotherapy was limited to neoadjuvant or conversion therapy；
8. Patients must have the ability to understand and voluntarily sign the informed consent, and must sign an informed consent before starting any specific procedure for the study；
9. Patients were considered capable of complying with the study protocol；
10. No medical comorbidities that could interfere with chemotherapy and immunotherapy or targeted therapy, see exclusion criteria；
11. Pre-treatment tumour tissue sample (if available). If tumour tissue is available, submit one formalin-fixed, paraffin-embedded (FFPE) tumour sample from a paraffin block (preferred), or approximately 10-15 slides containing unstained, freshly cut, serial sections, along with a relevant pathology report within 4 weeks of enrollment. If the FFPE samples described above are not available, any type of sample (including fine needle aspiration biopsy samples, cell mass samples [e.g., samples from pleural effusion] and lavage samples) may also be accepted. An associated pathology report should be provided with the sample. If tumour tissue is not available (e.g., exhausted due to past diagnostic tests), subjects are still eligible for study participation;
12. Adequate haematological and organ function， based on the following laboratory results obtained during the 14 days prior to enrollment (unless otherwise stated) ： Absolute neutrophil count (ANC)≥1.5×10 9 /L (1500/μL)， without supported granulocyte colony-stimulating factor Lymphocyte count ≥0.5×10 9 /L (500/μL) Platelets ≥ 75 × 10 9 /L（75, 000/μL） Haemoglobin≥ 85 g/L, blood transfusions may be permitted to meet this criterion Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 5 × upper limit of normal (ULN); Serum bilirubin≤ 3 × ULN Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥50 mL/min (using Cockcroft-Gault formula) Serum albumin≥28 g/L（2.8 g/dL） INR or aPTT≤2 × ULN, or PT prolonged ≤ 3 s if patients did not receive anticoagulant therapy.

    Albuminuria < 2+ tested by urinary cellulose (carried out within 14 days prior to initiation of treatment); Patients with baseline albuminuria ≥2+ should have their urine collected for 24 hours and must then confirm that albuminuria content within 24 hours is < 1g.
13. Any acute, clinically significant treatment-related toxicity (due to prior treatment) must have resolved to ≤ grade 1 prior to enrollment, except for hair loss;
14. HIV antibody test results were negative at screening;
15. Patients with active hepatitis B virus (HBV) infection: HBVDNA < 2000IU/mL acquired within 28 days prior to enrollment, receiving anti-HBV therapy (in accordance with local standard care, such as Entecavir) for at least 7 days prior to enrollment and willing to continue treatment during the study period; Patients with active hepatitis C virus (HCV) infection: HCVRNA < 2000IU/mL acquired within 28 days prior to enrollment, receiving anti-HCV therapy for at least 7 days prior to enrollment and willing to continue treatment during the study;
16. Women of childbearing age must undergo a negative pregnancy test (βHCG) before treatment, and women of childbearing age and men (who have sex with women of childbearing age) must agree to use effective contraception uninterrupted during treatment and for six months after the last therapeutic dose was administered.

Exclusion Criteria:

1. Colorectal cancer with extrahepatic metastasis;
2. Malignant abdominal effusion;
3. There were postoperative complications such as abdominal effusion, pleural effusion, intestinal cavity perforation, bleeding and intestinal obstruction that needed treatment.
4. History of soft meningitis
5. Current or past autoimmune diseases or immunodeficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granuloma, Sjogren's syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions: Subjects who had a history of autoimmune-related hypothyroidism and were receiving thyroid hormone replacement therapy were eligible; Subjects with controlled type 1 diabetes receiving insulin therapy were eligible; Subjects with clinical manifestations of eczema, psoriasis, chronic lichenia simple, or vitiligo only (e.g., excluding subjects with psoriatic arthritis) are eligible if they meet all of the following criteria: 1. Skin rash area must be < 10% body surface area 2. Good disease control at baseline with only inefficient topical glucocorticoid therapy. 3. No acute exacerbations requiring psoralen plus A-band ultraviolet radiation, methotrexate, retinoic acid, biologics, oral calcineurin inhibitors, or high-performance or oral glucocorticoid therapy have occurred in the previous 12 months;
6. Idiopathic pulmonary fibrosis, institutionalized pneumonia (e.g., bronchiolitis obliterans), drug-induced or idiopathic pneumonia, or evidence of active pneumonia on a chest computed tomography (CT) scan during screening. Radiation pneumonia was present in the allowable area (fibrosis)
7. Active TB disease
8. Major cardiovascular disease (such as New York Heart Society Class II or worse heart disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina in the 3 months prior to enrollment;
9. A history of congenital long QT syndrome or a corrected QT interval >500ms at screening (calculated using Fridericia's method);
10. A history of uncorrected electrolyte disturbances such as serum potassium, calcium, or magnesium
11. Received major surgery within 4 weeks prior to the enrollment (except for diagnosis) or expected to require major surgery during the study period;
12. Malignancies other than CRC that have developed within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, duct carcinoma in situ, or stage I uterine cancer;
13. Severe infections, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications, occurred in the 4 weeks prior to the enrollment;
14. Therapeutic antibiotics were given orally or intravenously within 2 weeks prior to the enrollment. Subjects who received prophylactic antibiotics (for example, to prevent urinary tract infections or exacerbations of COPD) were eligible;
15. Previous allogeneic stem cell or solid organ transplantation;
16. Received live attenuated vaccine within 4 weeks prior to the enrollment, or expected to receive such vaccine during sintilimab treatment or within 5 months after the last dose;
17. With untreated or incompletely treated esophageal and/or gastric varicose veins associated with bleeding or at high risk of bleeding. Prior to enrollment, subjects must undergo ultrasound, CT, MRI, or liver elasticity tests, assess the size of all varicose veins (small to large), and be treated according to local standard care. Subjects who received the corresponding examination within 6 months prior to the enrollment do not need to be re-examined;
18. Co-infection with HBV and HCV. Subjects with a history of HCV infection but negative PCR results for HCV RNA are considered not infected with HCV;
19. Symptomatic, untreated, or progressive central nervous system (CNS) metastases. Asymptomatic subjects whose CNS lesions have been treated are eligible as long as they meet all of the following criteria: They must have measurable lesions outside the CNS according to RECIST v1.1; Subjects had no history of intracranial or spinal bleeding; Metastases are limited to the cerebellar or supratentorial regions (i.e., no midbrain, pontine, medullary, or spinal cord metastases); No evidence of progress between completion of CNS oriented therapy and initiation of study therapy; Subjects had not received stereotactic, whole brain radiation, and/or neurosurgical resection within 28 days prior to the enrollment; There was no need for continuous use of glucocorticoids to treat CNS disease. A steady dose of anticonvulsant therapy is permitted. Asymptomatic subjects with newly detected CNS metastases at the time of screening are eligible after radiotherapy or surgery, and no need for repeated screening of brain scan results;
20. Refuse follow-up and participating in other clinical trials that may interfere with this study;
21. Patients are not suitable for enrollment judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival rate (1-year RFS) | 12 months
  Incidence of recurrence-free patients in one year

SECONDARY OUTCOMES:
recurrence-free survival (RFS) | Up to approximately 2 years
  time from surgery to recurrence or death
overall survival (OS) | Up to approximately 5 years
  time from enrollment to death
Safety and tolerability | Up to approximately 2 years
  adverse effect，Incidence of Adverse Events and Treatment-Emergent Adverse Events [Safety and Tolerability]
health-related quality of life (HRQol) | Up to approximately 2 years
  using patient-reported outcomes(PROs) via The European Organisation for Research and Treatment of Cancer(EORTC) Quality of Life Questionnaire Core 30 items (QLQ-C30)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No